CLINICAL TRIAL: NCT05650710
Title: Intraoperative Identification and Stimulation of the Ansa Cervicalis Nerve Plexus
Brief Title: Intraoperative Ansa Cervicalis Nerve (ACN) Stimulation
Acronym: ACS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, David Kent, Associate Professor, Department of Otolaryngology-Head and Neck Surgery, Vanderbilt University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 221998
Record Dates: First submitted 2022-12-06; First posted 2022-12-14 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Cancer; Obstructive Sleep Apnea
MeSH Terms: conditions — Head and Neck Neoplasms; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: All patients who meet eligibility will undergo uni- or bilateral neck dissection and other indicated procedures for management of head and neck cancer and will have measurements and photos/videos of the common trunks taken. An electrode will be placed on one or both common trunks to stimulate infrahyoid muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Surgical Procedure (Other): Consented patients who meet eligibility will have a surgical procedure for management of head and neck cancer, with dissection and exposure of the relevant anatomic structures as part of regular clinical care.
  Interventions: Device: Nerve stimulation using nerve stimulation device and sterile wire electrode.

INTERVENTIONS:
Device: Nerve stimulation using nerve stimulation device and sterile wire electrode. — A nerve stimulator device will be used in this study as a research tool to investigate whether a future (currently nonexistent) medical device might be able to stimulate desired infrahyoid musculature in a therapeutic manner.

SUMMARY:
Recently published data suggest that stimulation of the infrahyoid strap muscles increases pharyngeal patency in patients with obstructive sleep apnea, but the innervation of these muscles by the ansa cervicalis is variable. The investigators propose a study examining the anatomic variation of the ansa cervicalis and the effect of neurostimulation on muscle recruitment.

DETAILED DESCRIPTION:
This is a single-arm physiology study. Consenting patients undergoing neck dissection (ND) for cervical lymphadenectomy of level IV will undergo dissection of the ansa cervicalis nerves to the infrahyoid strap muscles. Per routine care, a large incision is made across the neck to provide surgeons access to the cervical lymph nodes for extirpation. During this dissection, the branch(es) of the ansa cervicalis nerve plexus descending from the loop of the plexus and innervating the infrahyoid strap muscles (the "common trunk") are dissected uni- or bilaterally. For this study, measurements and photos/videos of the common trunks will be taken. An electrode will be placed on one or both common trunks to stimulate infrahyoid muscles.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years old).
* Scheduled for uni- or bilateral neck dissection (BND) for cervical lymphadenectomy of level IV and other indicated procedures for management of head and neck cancer.

Exclusion Criteria:

* Unable to consent for research due to a pre-existing neurologic condition as determined by PI.
* Unable to consent for research due to language barriers.
* History of prior neck surgery with transection of the infrahyoid strap muscles as determined by clinical history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Primary Objective | Collected during a single operative procedure, taking about 15 minutes
  Anatomic measurements of the length, diameter, and comformation of the common trunk of the ansa cervicalis to the sternothyroid muscle and it's dependent branches, measured in mm with a flexible ruler.

SECONDARY OUTCOMES:
Secondary Objective | Collected during a single operative procedure, taking about 15 minutes.
  The amount of caudal movement of the thyroid cartilage and hyoid bone with stimulation of the common trunk of the ansa cervicalis to the sternothyroid muscle and it's dependent branches, measured in mm with a flexible ruler.
Secondary Objective | Collected during a single operative procedure, taking about 15 minutes.
  Anatomic confirmation of the common trunk of the ansa cervicalis to the sternothyroid muscle and it's dependent branches, documented with photography.

CONTACTS AND LOCATIONS:
Overall Officials: David T. Kent, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No